CLINICAL TRIAL: NCT04172545
Title: Impact of Anesthetic Conditions on Stapling Quality Measured as Staple Thickness During Laparoscopic Sleeve Gastrectomy
Brief Title: Observational Study on Effect of Anesthetic Conditions on Stapling Thickness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Prof Dr, AZ Sint-Jan AV
Other Study IDs: 2020OSstaplingcondition
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: stapling — staples are fired through the gastric wall after waiting several seconds for compression without attention to blood pressure, fluids given or intra abdominal pressure, but these might have an impact on quality of stapling. therefore the conditions during stapling will be recorded during stapling.

SUMMARY:
Measure anesthetic condition used during laparoscopic sleeve gastrectomy stapling. Measure quality of stapling in resected stomach by measuring staple thickness. Find if any relation exists.

DETAILED DESCRIPTION:
During each staple firing the staple size, time of compression and anesthetic conditions being systolic arterial pressure, fluids transfused and intra abdominal pressure used are recorded.

After removal of stapled stomach during surgery, thickness of stomach wall and thickness of staple line are measured and compared to evaluate quality of staple formation.

the closer the staple height to the wall thickness the better the quality of stapling. Because no one has ever analyzed this relationship, and certainly not under different anesthetic conditions it is not clear yet if any relationship will be found.

the analysis will help to understand the relation and help to start perhaps a randomised trial to learn what conditions are best to improve staple quality.

ELIGIBILITY:
Inclusion Criteria:

* primary sleeve gastrectomy

Exclusion Criteria:

* stomach disease
* prior surgery on the stomach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients undergoing bariatric surgery for the first time and where a sleeve gastrectomy is performed.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
thickness of staple line | intra operative on excised stomach before being discarded
  thickness of staple line measured in micrometers

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No